CLINICAL TRIAL: NCT05918744
Title: Sleep Extension and Vascular Health Study
Brief Title: Sleep and Vascular Health Study
Acronym: SAVHS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Auburn University (Other)
Responsible Party: Principal Investigator, Austin Robinson, Assistant Professor, Auburn University
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: AU IRB #23-172
Record Dates: First submitted 2023-06-08; First posted 2023-06-26 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Sleep; Vascular Diseases; Metabolic Disease
MeSH Terms: conditions — Vascular Diseases; Metabolic Diseases

STUDY DESIGN:
Intervention Model Description: Participants will serve as their own controls. Due to the nature of the intervention (extending time in bed by 1 hour) all participants will be measured in their habitual sleep state followed by their extended sleep state.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Habitual Sleep (No Intervention): Participants will follow their normal sleep schedule for 2 weeks.
- Sleep extension (Experimental): Participants will extend their time in bed by one hour for 2 weeks while being monitored.
  Interventions: Behavioral: Sleep Extension

INTERVENTIONS:
Behavioral: Sleep Extension — Participants will extend their time in bed by one hour for 2 weeks while being monitored.
  Arms: Sleep extension

SUMMARY:
Habitual short sleep duration (< 7 hours/night) increases the risk of cardiovascular disease (CVD) and all-cause mortality. Yet most adults, especially emerging adults (i.e., 18-25 years) do not achieve the National Sleep Foundation recommendation of 7-9 hours of sleep each night. Additionally, the American Heart Association recently included sleep duration in the "Life's Essential 8". This recent development emphasizes the importance of sleep and the need to advance our understanding of how sleep impacts cardiometabolic health (CMH), particularly in emerging adults, a population whose CVD risk trajectory is malleable. Specifically, emerging adulthood is a critical age window when age-related loss of CMH accelerates. Based on my previous work and others, both self-reported and objective measures of poor sleep (e.g., duration, variability) are linked to early signs of elevated CVD risk in emerging adults, such as microvascular dysfunction and elevated central blood pressure (BP), which precede the development of hypertension.

DETAILED DESCRIPTION:
The investigators aim to address the knowledge gap on whether sleep extension is a viable strategy to improve CMH in emerging adults with habitual short sleep duration. A prior study demonstrated the feasibility of sleep extension to improve BP and perceived sleepiness in predominantly normotensive emerging adults (18-23 years). Even without hypertension, reductions in BP are generally beneficial for CMH. The research hypothesis is that sleep extension (one extra hour in bed per night) will improve CMH and health behaviors in emerging adults who self-report < 7 hours of sleep per night. The primary aim is to determine if sleep extension is effective in improving BP. Investigators will assess CMH after habitual sleep (2 weeks) followed by a 2-week sleep extension intervention in 60 emerging adults (~30 female).

ELIGIBILITY:
Inclusion Criteria:

* 18 - 25 years old
* self-report sleeping less than 7 hours a night on average
* free from metabolic disease
* free from liver disease
* free from pulmonary disease
* free from cardiovascular disease

Exclusion Criteria:

* blood pressure higher than 140/80 mmHg
* BMI greater than 35 kg/m2
* use of blood thinners
* history of sleeping disorders
* no severe food allergies or eating disorders

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2025-05-05 (Estimated)

PRIMARY OUTCOMES:
Blood pressure reactivity | Change score from habitual sleep to day 15 (after 14 days of sleep extension)
  The investigators will measure blood pressure using photoplethysmography at the finger during rest and handgrip exercise.
Passive Leg movement | Change score from habitual sleep to day 15 (after 14 days of sleep extension)
  Passive leg movement will be used assessed blood flow responses to movement. The investigators will usie continuous measures of femoral artery diameter and velocity via duplex Doppler ultrasound (Hitachi Arietta 70) to calculate blood flow at rest and with the passive lelg movement. The femoral artery will be imaged in the longitudinal plane distal to the inguinal crease using a high-frequency (10-12 MHz) linear-array probe.
  Participants will be in a seated, reclined position with the lower leg free hanging. The ultrasound probe will be positioned by a lab member and the image will be recorded throughout triplicate 60-s measurements. Another lab member will independently move the lower leg through 90º range of motion at a rate of 1 Hz.
Circulating intercellular adhesion molecule 1 (ICAM-1) | Change score from habitual sleep to day 15 (after 14 days of sleep extension)
  Researchers will assess circulating markers intercellular adhesion molecule 1 (ICAM-1) using ELISA; samples will be run in triplicate and with quality controls.
Circulating Vascular adhesion molecule 1 (VCAM-1) | Change score from habitual sleep to day 15 (after 14 days of sleep extension)
  VCAM-1 will be assessed using ELISA ; samples will be run in triplicate and with quality controls
Objective sleep duration | Change score from habitual sleep to day 15 (after 14 days of sleep extension)
  Philips actiwatch spectrum will be used to quantify sleep duration. Participants will wear the watch units for 14 days. The investigators will assess sleep duration and cross-check actigraphy wear times with a sleep diary.
Objective sleep efficiency | Change score from habitual sleep to day 15 (after 14 days of sleep extension)
  Philips actiwatch spectrum will be used to quantify % of time in bed actually spent sleeping to calculate sleep efficiency.
Subjective sleep duration | Change score from habitual sleep to day 15 (after 14 days of sleep extension)
  The investigators will use the Pittsburgh Sleep Quality Index to asses sleep duration reflective of the one month period leading into the study.
Subjective sleep quality | Change score from habitual sleep to day 15 (after 14 days of sleep extension)
  The investigators will use the Pittsburgh Sleep Quality Index to assess perceived sleep quality reflective of the one month period leading into the study. The global score scale is 0 to 21.
Subjective Sleepiness | Change score from habitual sleep to day 15 (after 14 days of sleep extension)
  The investigators will administer the Epworth Sleepiness Scale (ESS). The scale is scored as 0-10 (normal sleepiness), 11- 14 (mild sleepiness), 15-17 (moderate sleepiness), and 18 -24 (severe sleepiness).
Pulse wave analysis | Change score from habitual sleep to day 15 (after 14 days of sleep extension)
  The investigators will use the SphygmoCor XCEL system to assess pulse wave analysis (PWA) The sampling site is the brachial artery (upper alarm instrumented with a cuff for oscillometric sphygmomanometer). PWA will be expressed as % (calculated as augmentation pressure divided by the pulse pressure).
Pulse wave velocity | Change score from habitual sleep to day 15 (after 14 days of sleep extension)
  The investigators will use the SphygmoCor XCEL system to assess pulse wave velocity (PWV) The sampling site is the carotid artery (tonometry) and femoral artery (upper leg instrumented with a cuff for oscillometric sphygmomanometer). PWW will be expressed as meters per second.
Cognitive motor task | Change score from habitual sleep to day 15 (after 14 days of sleep extension)
  The investigators will use a dual task assessment that involves walking an responding to prompts.
Circulating Leptin | Change score from habitual sleep to day 15 (after 14 days of sleep extension)
  Blood sample will be analyses with an enzyme-linked immunosorbent assay (ELISA) kit.
Circulating Ghrelin | Change score from habitual sleep to day 15 (after 14 days of sleep extension)
  Blood sample will be analysed with an enzyme-linked immunosorbent assay (ELISA) kit.

SECONDARY OUTCOMES:
Cardiorespiratory fitness | Pre- intervention
  The investigators will use indirect calorimetry to measure the participant's maximal oxygen consumption (VO2max) during incremental exercise on a treadmill. The investigators will use a Parvo TrueOne metabolic cart and Woodway treadmill.
Mental health - social anxiety | Change score from habitual sleep to day 15 (after 14 days of sleep extension)
  The investigators will administer the Liebowitz Social Anxiety Scale. The scale starts at 0 (none) and ends at 3 (severe) for 24 questions related to anxiety and avoidance, and a cumulative score is calculated.
Appetite Assessment | Change score from habitual sleep to day 15 (after 14 days of sleep extension)
  Appetite assessment via a visual analog scale (0 not feeling hungry/thirsty to 150 hungry/thirsty) and an ad libitum breakfast to measure food intake will take place during each of the experimental visits.
Hematocrit | Change score from habitual sleep to day 15 (after 14 days of sleep extension)
  Blood samples will be analyzed for hematocrit content (Thermo Hematocrit Microcentrifuge).
Hemoglobin | Change score from habitual sleep to day 15 (after 14 days of sleep extension)
  Blood samples will be analyzed for hemoglobin content (HemoCue, radiometer)
Urine Osmolarity | Change score from habitual sleep to day 15 (after 14 days of sleep extension)
  Researchers will analyze 24-hour urine samples for osmolarity (AI Osmometer 3D3)
Urine Electrolytes | Change score from habitual sleep to day 15 (after 14 days of sleep extension)
  Researchers will analyze 24-hour urine samples for electrolyte (Na, K, Cl) content using the SmartLyte Electrolyte Analyzer. The Na, K, Cl will be expressed as milliequivalents (mEq).
Blood Glucose | Change score from habitual sleep to day 15 (after 14 days of sleep extension)
  Researchers will analyze blood for glucose concentrations using the Cholestech.
Blood Cholesterol | Change score from habitual sleep to day 15 (after 14 days of sleep extension)
  Researchers will analyze blood for cholesterol (total, LDL and HDL) using the Cholestech.
Circulating Insulin | Change score from habitual sleep to day 15 (after 14 days of sleep extension)
  Blood sample will be analyses with an enzyme-linked immunosorbent assay (ELISA) kit.
Oxidized LDL | Change score from habitual sleep to day 15 (after 14 days of sleep extension)
  Blood sample will be analyses with an enzyme-linked immunosorbent assay (ELISA) kit.

CONTACTS AND LOCATIONS:
Locations (1):
- Auburn University, Auburn, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Grandner MA, Hale L, Moore M, Patel NP. Mortality associated with short sleep duration: The evidence, the possible mechanisms, and the future. Sleep Med Rev. 2010 Jun;14(3):191-203. doi: 10.1016/j.smrv.2009.07.006. Epub 2009 Nov 25. PMID 19932976
- [Background] Stock AA, Lee S, Nahmod NG, Chang AM. Effects of sleep extension on sleep duration, sleepiness, and blood pressure in college students. Sleep Health. 2020 Feb;6(1):32-39. doi: 10.1016/j.sleh.2019.10.003. Epub 2019 Nov 19. PMID 31753739
- [Background] Hirshkowitz M, Whiton K, Albert SM, Alessi C, Bruni O, DonCarlos L, Hazen N, Herman J, Katz ES, Kheirandish-Gozal L, Neubauer DN, O'Donnell AE, Ohayon M, Peever J, Rawding R, Sachdeva RC, Setters B, Vitiello MV, Ware JC, Adams Hillard PJ. National Sleep Foundation's sleep time duration recommendations: methodology and results summary. Sleep Health. 2015 Mar;1(1):40-43. doi: 10.1016/j.sleh.2014.12.010. Epub 2015 Jan 8. PMID 29073412
- [Background] Lloyd-Jones DM, Allen NB, Anderson CAM, Black T, Brewer LC, Foraker RE, Grandner MA, Lavretsky H, Perak AM, Sharma G, Rosamond W; American Heart Association. Life's Essential 8: Updating and Enhancing the American Heart Association's Construct of Cardiovascular Health: A Presidential Advisory From the American Heart Association. Circulation. 2022 Aug 2;146(5):e18-e43. doi: 10.1161/CIR.0000000000001078. Epub 2022 Jun 29. PMID 35766027
- [Background] Krefman AE, Labarthe D, Greenland P, Pool L, Aguayo L, Juonala M, Kahonen M, Lehtimaki T, Day RS, Bazzano L, Muggeo VMR, Van Horn L, Liu L, Webber LS, Pahkala K, Laitinen TT, Raitakari O, Lloyd-Jones DM, Allen NB. Influential Periods in Longitudinal Clinical Cardiovascular Health Scores. Am J Epidemiol. 2021 Nov 2;190(11):2384-2394. doi: 10.1093/aje/kwab149. PMID 34010956